CLINICAL TRIAL: NCT03594799
Title: Effects of a Nutritional Cocktail Consisting of Anti-oxidant and Anti-inflammatory Supplements to Prevent the Deconditioning Induced by 60 Days of Antiorthostatic Bed Rest
Brief Title: A New Nutritional Countermeasure to Prevent the Deconditioning Induced by 60 Days of Antiorthostatic Bed Rest
Acronym: LTBRCocktail
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre National d'Etudes Spatiales (Other Government)
Collaborators: European Space Agency (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 14-981
Record Dates: First submitted 2017-11-24; First posted 2018-07-20 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Weightlessness; Weightlessness; Adverse Effect
Keywords: Simulated Microgravity; Weightlessness; Countermeasure; Bedrest

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bed Rest Control Group (Experimental): 60 days of strict head-down tilt bed rest
  Interventions: Other: Bed Rest Control Group
- Cocktail intervention (Experimental): 60 days of strict head-down tilt bed rest along with a Cocktail supplementation composed of natural antioxidants XXS-2A-BR2 comprising vitamin E, Selenium and coupled with omega-3
  Interventions: Dietary Supplement: Cocktail intervention

INTERVENTIONS:
Other: Bed Rest Control Group — Subjects are in strict head down tilt bed rest at all time (including for taking showers etc.) for 60 days.
  Arms: Bed Rest Control Group
Dietary Supplement: Cocktail intervention — Subjects are in strict head down tilt bed rest at all time (including for taking showers etc.) for 60 days. In addition subjects are receiving a daily supplementation of a Cocktail. The daily dose of Cocktail consists of 6 pills per day: 2 at breakfast, 2 at lunch and 2 at diner. This will be equivalent to a daily dose of around 741 mg of bioactive polyphenols associated with Omega-3, Selenium and Vitamine E.
  Arms: Cocktail intervention

SUMMARY:
The objective of this study is to investigate whether the cocktail of natural antioxidants XXS-2A-BR2 comprising vitamin E and coupled with omega-3 helps to prevent and / or reduce the deleterious effects induced by long term physical inactivity through antiorthostatic bedrest. During a randomized 60 day bed rest study in 20 healthy male adults the two following aims will be undertaken:

* Sixteen scientific protocols will assess the changes in the cardiovascular, metabolism, muscle, bone, neuro sensorial, hematological and immunology systems.
* In the above mentioned systems, the potential beneficial effects of the countermeasure protocol will also be investigated.

DETAILED DESCRIPTION:
Space flights have shown the possibilities and limitations of human adaptation to space. For the last 50 years, results showed that the space environment and microgravity in particular, cause changes that may affect the performance of astronauts. These physiological changes particularly challenge the cardiovascular, metabolic, muscle and bone functions. Space agencies regularly conduct simulations on the ground on healthy volunteers to mimic the effects of weightlessness (head down bed rest model) to better understand the mechanisms of adaptations of the organism to space, and develop ways to prevent and / or reduce the negative biological effects of microgravity on astronauts. These protocols are called countermeasures. Since the beginning of space missions, various countermeasures have been tested on the ground and in-flight, including different exercise protocols. To date, however, none has been entirely satisfactory and space agencies continue to conduct simulation studies to evaluate new countermeasures. Nowadays, the human spaceflight program has entered the next phase of space exploration towards the Moon and Mars and there are clearly inherent medical challenges with such a goal, among which, countermeasure developments are a clear priority.

Based on recent evidences, the next countermeasure to be tested during a 60-day bed rest includes a nutritional countermeasure composed of an anti-oxidant and anti-inflammatory dietary mix.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteer (see below the description of medical tests and laboratory analysis performed at the selection visit),
* Age 20 to 45,
* No overweight nor excessive thinness with BMI (weight Kg/ height m2) between 22 and 27,
* Height between 158 and 190 cm,
* No personal nor family past record of chronic or acute disease or psychological disturbances which could affect the physiological data and/or create a risk for the subject during the experiment,
* Fitness level assessment:

  * if age < 35 years: 35 ml/min./kg < VO2max < 60ml/min./kg,
  * if age > 35 years: 30 ml/min./kg < VO2max < 60ml/min./kg
* Active and free from any orthopedic, musculoskeletal and cardiovascular disorders,
* Non smokers,
* No alcohol, no drug dependence and no medical treatment,
* No shift work or travel across more than one time zone in previous 2 months,
* Covered by a Social Security system,
* Have signed the information consent,
* Free of any engagement during the three hospitalization planned periods.

Exclusion Criteria:

* - Past record of orthostatic intolerance,
* Cardiac rhythm disorders,
* Chronic back pains,
* History of hiatus hernia or gastro-esophageal reflux,
* History of thyroid dysfunction, renal stones, diabetes, migraines,
* Past records of thrombophlebitis, family history of thrombosis or positive response in thrombosis screening procedure,
* Allergy including xylocaine allergy
* Abnormal result for lower limbs echo-doppler,
* History or active claustrophobia,
* History of genetic muscle and bone diseases of any kind,
* History of sleep disorders, no shift work or travel across more than one time zone in previous two months
* Vestibular disorders,
* Audition problem,
* Vision corrected no more than 20/30, color-blindness
* Bone mineral density: T-score ≤ -1.5,
* Osteosynthesis material, presence of metallic implants,
* History of knee problems or joint surgery/broken leg
* Poor tolerance to blood sampling,
* Having given blood (more than 8ml/kg) in a period of 8 weeks or less before the start of the experiment,
* Special food diet, vegetarian or vegan, food allergy especially allergic to peanut or soya.
* Positive reaction to any of the following tests: HVA IgM (hepatitis A), HBs antigen (hepatitis B), anti-HVC antibodies (hepatitis C), anti-HIV1+2 antibodies,
* Subject already participating or in the exclusion period of a clinical research,
* Refusal to give permission to contact his general practitioner,
* Incarcerated persons,
* Subject who, in the judgment of the investigator, is likely to be non-compliant during the study, or unable to cooperate because of a language problem or poor mental development,
* Subject who has received more than 4500 Euros within 12 months for being a research subject.
* Subject under guardianship or trusteeship.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Change in fasting plasma triglycerides concentration | 60 days
  Plasma triglycerides concentration will be analyzed by enzymatic colorimetric method (reagent kit) after ultracentrifugation to isolate chylomicrons and Very Low Density Lipoproteins

SECONDARY OUTCOMES:
Change in vertebral bone marrow fat fraction. | 60 days
  This will be performed by using MR scanning sequences that specifically measure water and fat signals then calculate the respective content.
Change in B lymphopoiesis | 60 days
  Next generation sequencing (NGS) of IgM heavy chain transcripts extracted from PBMC will 1) indicate if the expression frequencies of Ig gene segments are modified during bed rest thereby indicating a change in B lymphopoiesis (because each B cell created in the marrow is characterized by its own VH-D-JH-Cµ mRNA) and 2) allow the assessment of the activities of enzymes required for the formation of the B cell antigen receptor repertoire.
  Flow cytometry will be used to determine if there is an egress of HSC/progenitors from the bone marrow into blood stream thereby indicating a decrease of the interactions between HSC and their niche. The same technique will be used to determine if there are changes in B cell subsets in peripheral blood.
Changes in myokines. | 60 days
  Mass spectrometry will be performed on proteins obtained from muscle biopsies, microdialysis and serum. The generated peptides will be analysed using high resolution mass shot-gun mass spectrometry.
Change in cardio-postural stability | 60 days
  The end point is a reduction in muscle pump indices: a) decrease in causality between EMG and Blood pressure, b) decrease in gain between EMG and Blood pressure, and c) decrease in the interaction time between EMG and Blood pressure.
Change in insulin sensitivity | 60 days
  Skeletal muscle insulin resistance will be assessed during a euglycaemic hyperinsulinaemic clamp.
  Whole blood will be immediately analyzed for glucose concentration, serum insulin will be quantified by radioimmunoassay and catecholamines will be quantified by high-performance liquid chromatography. Peripheral insulin sensitivity will be calculated during the final hour of the clamp in steady state.
Changes in brain structure | 60 days
  Both structural and functional brain changes associated with head-down bedrest will be examined by 3T MRI. Imaging sequence parameters will be selected to maximize sensitivity to effects of interest.
Change in head movements in response to a virtual projectile | 60 days
  Subjects perform a video game-like task of shooting a projectile out of a hand-held tool so that it passes between the gaps of an oriented target grill. Since the projectile and the tool are long and narrow, the subject must place the tool at the same orientation as the grill to achieve success. On certain trials, the subject is required to move the head between the time that the target is acquired and the moment of the response. Trials vary in terms of what the subject can see and feel during the execution of the task, and on body posture.
  A 3D motion caption system is used to track in real-time the movements of the subject' head and hands. A virtual reality helmet is used to provide visual and audio information. A moving head support will be used to allow the subject to tilt the head laterally in both seated and laying conditions.
Change in pulse wave velocity in carotid and femoral arteries | 60 days
  Change in pulse wave velocity in carotid and femoral arteries will be assessed by non-invasive ultrasound measurements.
Adipose Tissue Transcriptomics | 60 days (pre and post bed rest)
  Within-subjects changes in adipose gene expression between intervention groups will be evaluated using RNAseq
Measurement of changes to the sleep electroencephalogram (EEG) | 60 days
  Measurement of changes to objective sleep will be determined using continuous 24-h EEG monitoring at regular intervals throughout the protocol (including baseline, head down tilt, and recovery).
Measurement of changes in subjective sleep quality | 60 days
  Changes in subjective sleep quality will be measured using the Karolinska sleepiness scale (KSS) four times per day (mealtimes and bed time) doing every day of the protocol.
Measurement of changes in circadian rhythms of melatonin and cortisol | 60 days
  Changes to the circadian rhythms of melatonin and cortisol will be measured by radioimmunoassay on saliva samples taken hourly throughout the day at regular intervals throughout the protocol (including baseline, head down tilt, and recovery; same as for EEG).
Measurement of changes in the whole-blood transcriptome in response to 60-day head down tilt bed rest | 60 days
  Changes to the circadian rhythmicity of the whole-blood transcriptome will be measured by whole-genome microarray analyses of RNA extracted from six 4-hourly blood samples taken over a 24-h period at regular intervals throughout the protocol (including baseline, head down tilt, and recovery; same as for EEG).
Change in levels of S-nitrosylated proteins | 60 days
  Vastus Lateralis needle biopsies will be performed before, at the end of the Head Down Tilt period (after about 60 days of bedrest) and of the recovery phases. Change in levels of S-nitrosylated proteins will be measured in active vs. atrophic muscle following extended bed rest.
Change in skeletal muscle gene expression (transcriptome) | 60 days
  Vastus Lateralis needle biopsies will be performed before, at the end of the Head Down Tilt period (after about 60 days of bedrest) and of the recovery phases. Change in skeletal muscle gene expression will be analyzed by microarray technology.
Change in bone resorption marker CTX | 60 days
  Bone resorption marker CTX will be analyzed in the aliquots of total 24h-urine, collected at different timepoints of the study (pre, during and after the bedrest phase).
Change in de novo lipogenesis | 60 days
  Energy substrates labeled with stable (non radioactive) isotopes will be used to measure intermediary metabolism and fluxes.
Accuracy and precision of vestibular-evoked sway responses | 60 days
  In a healthy standing subject, Galvanic Vestibular Stimulation (GVS) evokes a postural sway response directed towards the anode electrode. The direction of the response is fixed in head coordinates and so it will rotate as the head is turned. To determine if bedrest has affected the accuracy and precision of this sway response, we will measure the direction of the ground reaction force (GRF) response evoked by GVS in standing volunteers under different head orientations. The mean direction (accuracy) along with the trial-to-trial variability (precision) of the GRF vector will be separately determined. Any reduction in accuracy or precision will indicate degraded vestibular control of balance.
Change in T wave morphology | 60 days
  24h ECG Holters will be done at different timepoints of the study (pre, during and after the bedrest phase). A conventional Holter analysis will be performed using dedicated commercial software. Moreover, the recordings obtained will be analyzed using several advanced signal processing techniques, which will be focused on different aspects of ventricular repolarization.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud BECK, MD, Principal Investigator — MEDES - IMPS
Locations (1):
- Medes-Imps, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trim WV, Walhin JP, Koumanov F, Turner JE, Shur NF, Simpson EJ, Macdonald IA, Greenhaff PL, Thompson D. The impact of physical inactivity on glucose homeostasis when diet is adjusted to maintain energy balance in healthy, young males. Clin Nutr. 2023 Apr;42(4):532-540. doi: 10.1016/j.clnu.2023.02.006. Epub 2023 Feb 16. PMID 36857962
- [Derived] Stratis D, Trudel G, Rocheleau L, Pelchat M, Laneuville O. The Characteristic Response of the Human Leukocyte Transcriptome to 60 Days of Bed Rest and to Reambulation. Med Sci Sports Exerc. 2023 Mar 1;55(3):365-375. doi: 10.1249/MSS.0000000000003071. Epub 2022 Oct 15. PMID 36251376
- [Derived] Trim WV, Walhin JP, Koumanov F, Bouloumie A, Lindsay MA, Travers RL, Turner JE, Thompson D. The Impact of Long-term Physical Inactivity on Adipose Tissue Immunometabolism. J Clin Endocrinol Metab. 2022 Jan 1;107(1):177-191. doi: 10.1210/clinem/dgab647. PMID 34480570
- [Derived] Austermann K, Baecker N, Zwart SR, Fimmers R, Frippiat JP, Stehle P, Smith SM, Heer M. Antioxidant Supplementation Does Not Affect Bone Turnover Markers During 60 Days of 6 degrees Head-Down Tilt Bed Rest: Results from an Exploratory Randomized Controlled Trial. J Nutr. 2021 Jun 1;151(6):1527-1538. doi: 10.1093/jn/nxab036. PMID 33831949
- [Derived] Liu T, Melkus G, Ramsay T, Sheikh A, Laneuville O, Trudel G. Bone Marrow Reconversion With Reambulation: A Prospective Clinical Trial. Invest Radiol. 2021 Apr 1;56(4):215-223. doi: 10.1097/RLI.0000000000000730. PMID 33038096